CLINICAL TRIAL: NCT05736484
Title: The MOVE ON Trial: A Randomized Trial of Gamification and Coaching to Improve Mobility After Hospitalization
Brief Title: Randomized Clinical Trial to Improve Mobility After Hospitalization
Acronym: MOVE_ON
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 852338
Record Dates: First submitted 2023-02-06; First posted 2023-02-21 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Hypertension; Diabetes; Heart Failure; Ambulatory Difficulty; Mobility Limitation
Keywords: Gamification; Physical Activity; Behavioral Economics; Social Support; Mobility
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Heart Failure; Mobility Limitation; Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a 2-arm randomized control trial over 26 weeks with 26 weeks follow-up (total of 52 weeks) that compares a control group wearing a wearable activity tracker to the intervention group that uses the same device and receives a supportive social incentive-based gamification intervention.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants will receive a wearable device (e.g. FitBit) but no other interventions during the intervention or follow-up periods.Participants will complete milestones within the study, such as the Function assessment during the 6, and 12-month timepoints in the study. They will also complete a series of surveys during the 3, 6, 9, and 12-month timepoints in the study. Participants will complete an end-of-study questionnaire on their experience with the wearable device and time in the study.
- Social Support Gamification (Experimental): Intervention participants will receive a wearable device (e.g. FitBit) and will enter a game designed with behavioral economics concepts to address predictable barriers to behavior change during a 26-week intervention period. Participants will also work with a virtual health coach throughout the intervention period to increase their physical activity.
  At the end of the 26 week intervention period, participants will enter a 26 week follow-up period during which interventions will cease but passive data collection of step counts will continue. Participants will also complete milestones within the study, such as the Function assessment during the 6, and 12-month timepoints in the study. They will also complete a series of surveys during the 3, 6, 9, and 12-month timepoints in the study. Participants will complete an end-of-study questionnaire on their experience with the wearable device and time in the study.
  Interventions: Behavioral: Social Support Gamification

INTERVENTIONS:
Behavioral: Social Support Gamification — Participants sign a pre-commitment contract agreeing to try their best to achieve their daily step goal. Over the 26-week intervention period, participants are endowed 70 points (10/day) weekly and informed they will lose 10 points each day goal is not met. Points are replenished at start of each week. At the end of each week, if the participant has 40 points or more, they will advance a level, or drop a level if they have less than 40 points. The levels include blue (lowest), bronze, silver, gold, platinum (highest). Participants select a family member or friend as a support partner to receive weekly email on participants' progress (points, game level, and average step count). Participants will also work with a virtual health coach by attending group sessions organized by them with other participants through video calls once a month to discuss ways to motivate participants to increase their physical activity.
  Arms: Social Support Gamification

SUMMARY:
The objective of this study is to test the feasibility of using behavioral economic interventions (gamification with social incentives) to increase physical activity after hospital discharge to reduce incident mobility disability among older adults.

DETAILED DESCRIPTION:
MOVE ON is a 2-arm, randomized trial enrolling older adults 50 years or older with a recent hospitalization for hypertension, diabetes, and mild-moderate heart failure. The 52 week trial compares a control group wearing a wearable activity tracker to the intervention group that uses the same device and receives a supportive social incentive-based gamification intervention. The primary goal is to increase physical activity after discharge from the hospital to reduce incident mobility disability associated with acute illness and to reduce acute and post-acute care utilization.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years or older
* Admitted to the University of Pennsylvania Health System acute care hospital (Hospital of the University of Pennsylvania, Penn Presbyterian Medical Center, Pennsylvania Hospital, Lancaster General Health, Chester County Hospital, or Penn Medicine Princeton Medical Center) and discharged to home
* Able to ambulate independently

Exclusion Criteria:

* Inability to provide informed consent
* Does not have daily access to a smartphone compatible with the wearable device and is not willing to use a device that the investigators can provide participants' with
* Already enrolled in another physical activity study
* Low mobility score indicating that the patient is not able to walk distances greater than 1000 steps/day independently
* Any other medical conditions that would prohibit participation in a 6-month physical activity program
* Unable to complete the baseline period (must have at least 4 out of 7 days of step data with minimum step count of 1000 steps/day)
* Not willing to use the wearable device for the full duration of the study
* Enrolled in hospice

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in mean daily step count from baseline to the end of the 26 week intervention period. | Baseline to 26 week intervention period (Weeks 1-26)
  The primary outcome of the study is the participants' change in mean daily steps from the baseline period to the end of the 26 week intervention period collected by Fitbit Inspire device.

SECONDARY OUTCOMES:
Change in mean daily step count from baseline to the end of the 26 week follow-up period. | Baseline to 52 weeks- end of the study (Weeks 1-52)
  The secondary outcome will examine the change in participants' mean daily step counts from the baseline period to the end of the 26 week follow-up period after the end of the 26 week intervention period collected by the Fitbit device.
Participants' mobility disability throughout the entire study (Baseline to end of study [52 weeks]). | Baseline to 26 and 52 weeks- end of the study (Weeks 1-52)
  The investigators will explore participant mobility disability; defined as the change in the Patient-Reported Outcomes Measurement Information System (PROMIS) mobility measure score (on a scale of 5- without any difficulty to 1- unable to do) from baseline to 26 and 52 weeks, adjusting for time and participant baseline characteristics.
Participants' acute care utilization throughout the entire study (Baseline to end of study [52 weeks]). | Baseline to 26 and 52 weeks- end of the study (Weeks 1-52)
  The investigators will explore participants' acute care utilization; defined as the number of emergency department visits and hospitalizations that occur at 26 and 52 weeks, adjusting for time and participant baseline characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Greysen, MD, MHS, MA, Principal Investigator — University of Pennsylvania
Locations (1):
- Blockley Hall, Philadelphia, Pennsylvania, United States